CLINICAL TRIAL: NCT06033781
Title: Can a Brief Therapy Improve Pediatric Nightmares, Mental Health, and Suicidality?
Brief Title: Cognitive-Behavioral Therapy for Children With Nightmares
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oklahoma (Other)
Collaborators: University of Tulsa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15401
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Nightmare; Suicidal Ideation; Children, Only
Keywords: CBT; Cognitive; Behavioral; Therapy
MeSH Terms: conditions — Suicidal Ideation; Behavior | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Right-Away (Experimental): Child will start the CBT-NC treatment right away.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Nightmares in Children
- Waitlist Control (No Intervention): Waitlist control group will complete the assessments at the same time as the treatment group, without receiving any treatment. They will be offered treatment after finishing the waitlist.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Nightmares in Children — The Cognitive Behavioral Therapy for Nightmares in Children (CBT-NC) is a brief, five-session manualized therapy designed to treat children ages 6-17. The manualized CBT protocol is five session that teach sleep hygiene, relaxation strategies, and addresses nightmares therapeutically through exposure and rescripting.
  Arms: Treatment Right-Away

SUMMARY:
The goal of this clinical trial is to assess the efficacy of CBT-NC intervention to determine its impact on mental health and suicidality in children ages 6-17. The main aims are:

Aim 1: Examine CBT-NC efficacy for improving nightmare distress and frequency in youth with chronic nightmares by comparing the treatment and waitlist group.

Aim 2: Examine whether improvements in nightmares relate to fewer mental health problems for youth by determining by comparing the treatment and waitlist group.

DETAILED DESCRIPTION:
Chronic nightmares in youth put them at risk for mental health problems including suicidal ideation and attempts. Left untreated, chronic childhood nightmares can persist, resulting in myriad mental health problems. An international consortium of nightmare experts urged the medical community to prevent mental health problems in youth through early detection and treatment of chronic nightmares. There are several well-established, brief, and cost-effective nightmare treatments for adults but research with youth is lagging. To date, several small case series have investigated nightmare treatments for youth and there is a need for clinical trials. The proposed study will evaluate the efficacy of Cognitive Behavioral Therapy for Nightmares in Children (CBT-NC), a brief five-session manualized therapy designed to treat children ages 6-17. This randomized controlled trial with treatment and waitlist arms will assess the efficacy of the intervention and determine if the intervention has any impact on mental health problems and suicidality at follow-up.

This study will be the first randomized controlled trial to assess the efficacy of Cognitive behavioral therapy for nightmares in children (CBT-NC), compared to a waitlist group. Our goal is to determine whether CBT-NC can be an effective treatment strategy for reducing nightmares in youth, which are linked to suicidality.

First, this study will address the need for efficacious and cost-effective treatment for improving nightmare distress and frequency in youth with chronic nightmares. Second, this study will determine if improvements in nightmares reduce risk for youth mental health problems including suicidal ideation.

ELIGIBILITY:
Inclusion Criteria:

* Child must be between ages of 6-17 years 11 months.
* Child must report recurrent nightmares that meet Diagnostic and Statistical Manual of Mental Disorders criteria for nightmare disorder.
* Child must speak and understand English at no less than a 6-year-old level.
* Children on prescribed psychotropic medications must be stable for 30 days prior to enrolling.
* Child must have a parent or legal guardian attend study visits with them.
* Participants must have access to WIFI/phone data in order to participate in this study and must have an electronic device with a camera enabled.

Exclusion Criteria:

* Children with a diagnosis of sleep apnea which is not adequately treated.
* Children whose receptive/expressive language skills are below a 6-year-old level.
* If it is determined that a child is actively suicidal and at imminent risk for self-harm, the family will be notified and referred for immediate care. They will not be eligible for the study until they are deemed stable.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Changes in reports on Sleep Journal | Participants complete this daily from consent to baseline assessment (Week 0), during treatment, and before post-assessments, up to 20 weeks. They also complete a weekly version for 4 weeks following post-assessments (Weeks 10-14).
  The sleep journal is a 3 question self report regarding nightmares.
Change in Nightmare Disorder Diagnoses from Structure Clinical Interview for Sleep Disorders in Children (SCISD-Kid) | Participants will be assessed at baseline (Week 0) and at post-assessments, up to 20 weeks.
  The SCISD-Kid is a structured clinical interview that assesses for sleep disorders. The main module interest is the nightmare disorder module.
Change on the Columbia Suicide Severity Rating Scale (C-SSRS) | Participants will be assessed at baseline (Week 0), at post-assessments, up to 20 weeks, and weekly following their post-assessment for 4 weeks.
  The C-SSRS is a yes/no questionnaire to assess for suicidal ideations and behaviors. For this study, we will be looking at the 5 suicidal ideation questions.
Change on the Strengths and Difficulties Questionnaire (SDQ) - Caregiver Version | Participants' caregivers will be assessed at baseline (Week 0) and at post-assessments, up to 20 weeks.
  The SDQ is a 25-item brief behavioral screening questionnaire for detecting mental health problems in general populations people aged 2-17. It assesses three scales for internalizing problems (10 items), externalizing problems (10 items), and prosocial behavior (5 items). The internalizing and externalizing scales have scores ranging from 0 to 20 with higher scores indicating more difficulties. The prosocial behavior scale ranges from 0 to 10 with higher scores indicating more prosocial behaviors.
Change on the Patient Health-Questionnaire-9 (PHQ-9) | Participants will be assessed at baseline (Week 0) and at post-assessments, up to 20 weeks.
  The PHQ-9 is a 9-question Likert scale questionnaire to assess for depression. The items are scored on a scale of 0-27. Total scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe, and severe depression, respectively.

SECONDARY OUTCOMES:
Change on the Child Adolescent Trauma Screen (CATS) - Child Version | Participants will be assessed at baseline (Week 0) and at post-assessments, up to 20 weeks.
  The CATS screens for child trauma history and PTSD symptoms in youth ages 7-17; 15 YES/NO questions; 1 open-ended question
Change on the Patient Health-Questionnaire-2 (PHQ-2) | Participants will be assessed at baseline (Week 0), at post-assessments, up to 20 weeks, and weekly following their post-assessment for 4 weeks.
  The PHQ-9 is a 2-question Likert scale questionnaire to screen for depression. Scores range from 0-6. A score of 3 or greater indicates major depressive disorder may exist.
Change on the Child Adolescent Trauma Screen (CATS) - Caregiver Version | Participants' caregivers will be assessed at baseline (Week 0) and at post-assessments, up to 20 weeks.
  The CATS screens for child trauma history and PTSD symptoms in youth ages 7-17; 15 YES/NO questions; 1 open-ended question
Change on Sleep Locus of Control (SLOC) | Participants and caregivers will be assessed at Baseline (Week 0), post-assessments, and weekly during therapy, up to 20 weeks.
  The SLOC is a 5 item self report measure perceived contingencies between sleep behavior and events. This scale is collected as a child self report, and a caregiver report regarding child. The items are answered with a 1-5 Likert scale with total scores ranging from 5 to 25. Higher scores indicate higher locus of control.
Change on Nightmare Locus of Control (NLOC) | Participants and caregivers will be assessed at Baseline (Week 0), post-assessments, and weekly during therapy, up to 20 weeks.
  The NLOC is a 5 item self report measure regarding nightmare behavior and events. This scale is collected as a child self report, and a caregiver report regarding child. The items are answered with a 1-5 Likert scale with total scores ranging from 5 to 25. Higher scores indicate higher locus of control.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Cromer, PhD, Principal Investigator — University of Tulsa; Tara Buck, MD, Principal Investigator — University of Oklahoma
Locations (2):
- United States (2):
  - University of Tulsa, Tulsa, Oklahoma
  - University of Oklahoma School of Community Medicine, Tulsa, Oklahoma

IPD SHARING:
Plan to Share IPD: No